CLINICAL TRIAL: NCT02318329
Title: A Phase 1 Open-Label, Dose-Finding Study Evaluating Safety and Pharmacokinetics of FPA144 in Patients With Advanced Solid Tumors
Brief Title: Open-Label, Dose-Finding Study Evaluating Safety and PK of FPA144 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPA144-001
Record Dates: First submitted 2014-11-25; First posted 2014-12-17 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumors; Gastric Cancer; Transitional Cell Carcinoma of the Bladder
Keywords: FGFR2b, FGFR2, FGFR, bladder neoplasms, esophageal cancer
MeSH Terms: conditions — Stomach Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms | interventions — bemarituzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1A: FPA144 Dose Escalation Solid Tumors (Experimental): Dose escalation of FPA144 (0.3 mg/kg to 15 mg/kg)
  Interventions: Drug: FPA144
- Part 1B: FPA144 Dose Escalation Gastric Cancer (Experimental): Dose escalation of FPA144 (3-10 mg/kg) in patients with gastric cancer
  Interventions: Drug: FPA144
- Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors (Experimental): Evaluation of objective responses in patients with tumors with various levels of FGFR2b overexpression
  Interventions: Drug: FPA144

INTERVENTIONS:
Drug: FPA144 — FPA144 will be administered by IV infusion over approximately 30 minutes every 2 weeks.
  Other Names: Bemarituzumab

SUMMARY:
This is a three-part, open-label, safety, tolerability, and PK study of FPA144. Patients will be enrolled in Part 1 (A or B, dose escalation) or Part 2 (dose expansion) of the study, but not both.

DETAILED DESCRIPTION:
Part 1A is a dose-escalation study in patients with any locally advanced or metastatic solid tumor or lymphoma for which standard therapies have been exhausted. Part 1B will further assess safety and evaluate PK of FPA144 in gastric cancer patients.

Part 2 patients will be enrolled and treated in order to further characterize safety and preliminary efficacy in a selected cancer patient population with the greatest potential for clinical benefit from FPA144 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 3 months
* ECOG performance status of 0 to 1

  • In sexually-active patients, willingness to use 2 effective methods of contraception
* Adequate hematological and organ function, confirmed by lab values
* Tumor tissue must be available for prospective determination of FGFR2b overexpression

  * Locally recurrent or metastatic disease that has progressed on or following standard treatment, or is not a candidate for standard treatment
  * Histologically or cytologically confirmed transitional cell carcinoma of the genitourinary tract
  * Measurable disease as defined by RECIST version 1.1

Exclusion Criteria:

* Untreated or symptomatic central nervous system (CNS) metastases
* Impaired cardiac function or clinically significant cardiac disease

  - Treatment with any anticancer therapy or participation in another therapeutic clinical study with investigational drugs </=14 days (</=28 days for patients in Korea) prior to first dose of FPA144
* Ongoing acute adverse effects from prior anticancer or investigational therapy > NCI CTCAE Grade 1
* Retinal disease or a history of retinal disease or detachment
* Corneal defects, corneal ulcerations, keratitis, keratoconus, history of corneal transplant, or other known abnormalities of the cornea
* Major surgical procedures are not allowed ≤28 days prior to FPA144 administration
* Females who are pregnant or breastfeeding; women of childbearing potential must not be considering getting pregnant during the study

  - Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study
* Known allergy or hypersensitivity to components of the FPA144 formulation including polysorbate
* History of prior malignancy except:
* a) Curatively treated non-melanoma skin cancer or
* b) Solid tumor treated curatively more than 5 years previously without evidence of recurrence or
* c) History of other malignancy that in the Investigator's opinion would not affect the determination of study treatment effect
* Prior treatment with any selective inhibitor (e.g., AZD4547, BGJ398, JNJ-42756493, BAY1179470) of the FGF-FGFR pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-11; Primary Completion 2019-02-28 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Lead, Study Director — Five Prime Therapeutics, Inc.
Locations (26):
- United States (13):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, Mission Bay, San Francisco, California
  - Innovative Cancer Research Institute, Whittier, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Weill Cornell Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- South Korea (9):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be provided to investigative sites requesting information for secondary publication.
Supporting Information: Study Protocol
Time Frame: After publication of the primary endpoint results.
Access Criteria: Participating investigators in good standing.

REFERENCES:
- [Background] Catenacci DV, Tesfaye A, Tejani M, Cheung E, Eisenberg P, Scott AJ, Eng C, Hnatyszyn J, Marina N, Powers J, Wainberg Z. Bemarituzumab with modified FOLFOX6 for advanced FGFR2-positive gastroesophageal cancer: FIGHT Phase III study design. Future Oncol. 2019 Jun;15(18):2073-2082. doi: 10.2217/fon-2019-0141. Epub 2019 May 16. PMID 31094225
- [Background] Catenacci DVT, Rasco D, Lee J, Rha SY, Lee KW, Bang YJ, Bendell J, Enzinger P, Marina N, Xiang H, Deng W, Powers J, Wainberg ZA. Phase I Escalation and Expansion Study of Bemarituzumab (FPA144) in Patients With Advanced Solid Tumors and FGFR2b-Selected Gastroesophageal Adenocarcinoma. J Clin Oncol. 2020 Jul 20;38(21):2418-2426. doi: 10.1200/JCO.19.01834. Epub 2020 Mar 13. PMID 32167861
- [Background] Xiang H, Liu L, Gao Y, Ahene A, Macal M, Hsu AW, Dreiling L, Collins H. Population pharmacokinetic analysis of phase 1 bemarituzumab data to support phase 2 gastroesophageal adenocarcinoma FIGHT trial. Cancer Chemother Pharmacol. 2020 Nov;86(5):595-606. doi: 10.1007/s00280-020-04139-4. Epub 2020 Sep 23. PMID 32965540

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg: 3 + 3 dose escalation cohort with 0.3 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1A: FPA144 Dose Escalation Solid Tumors 1mg/kg: A traditional 3 + 3 dose escalation design will be implemented. Successive cohorts of patients (3/cohort) will each be started on a fixed dose of FPA144. Dose: 1.0 mg/kg FPA144 every 2 weeks in 28 day cycles for this cohort.
- Part 1A: FPA144 Dose Escalation Solid Tumors 3 mg/kg: A traditional 3 + 3 dose escalation design will be implemented. Successive cohorts of patients (3/cohort) will each be started on a fixed dose of FPA144. Dose: 3.0 mg/kg FPA144 every 2 weeks in 28 day cycles for this cohort.
- Part 1A: FPA144 Dose Escalation Solid Tumors 6 mg/kg: A traditional 3 + 3 dose escalation design will be implemented. Successive cohorts of patients (3/cohort) will each be started on a fixed dose of FPA144. Dose: 6.0 mg/kg FPA144 every 2 weeks in 28 day cycles for this cohort.
- Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg: A traditional 3 + 3 dose escalation design will be implemented. Successive cohorts of patients (3/cohort) will each be started on a fixed dose of FPA144. Dose: 10 mg/kg FPA144 every 2 weeks in 28 day cycles for this cohort.
- Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg: A traditional 3 + 3 dose escalation design will be implemented. Successive cohorts of patients (3/cohort) will each be started on a fixed dose of FPA144. Dose: 15 mg/kg FPA144 every 2 weeks in 28 day cycles for this cohort.
- Part 1B: FPA144 Dose Escalation Gastric Cancer 3 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 3.0 mg/kg IV every 2 weeks in 28 day cycles.
- Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg: Part 1B will be a 3 + 3 design and enroll patients with gastric cancer. Participants may be gastric cancer patients whose tumors will be tested retrospectively, or those who are known to be FGFR2 gene-amplified or FGFR2b protein-overexpressed. In a staggered fashion with Part 1A dose escalation, patients in Part 1B will be enrolled one dose level below the current highest dose level cohort being studied in Part 1A. Dose: 6.0 mg/kg FPA144 every 2 weeks in 28 day cycles for this cohort.
- Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg: Part 1B will be a 3 + 3 design and enroll patients with gastric cancer. Participants may be gastric cancer patients whose tumors will be tested retrospectively, or those who are known to be FGFR2 gene-amplified or FGFR2b protein-overexpressed. In a staggered fashion with Part 1A dose escalation, patients in Part 1B will be enrolled one dose level below the current highest dose level cohort being studied in Part 1A. Dose: 10 mg/kg FPA144 every 2 weeks in 28 day cycles for this cohort.
- Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors: Gastric and bladder cancer patients with tumors with FGFR2b overexpression administered FPA144 15mg/kg IV every 2 weeks in 28 day cycles. Dose established from prior dose escalation evaluation in parts 1A and 1B.
Period: Overall Study
Arm/Group | Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 1mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 6 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 3 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors
Started | 3 | 4 | 3 | 3 | 3 | 3 | 1 | 1 | 6 | 52
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 3 | 3 | 3 | 1 | 1 | 6 | 52
Not completed — Progressive Disease | 2 | 3 | 2 | 3 | 3 | 3 | 1 | 1 | 5 | 39
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Other | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients enrolled on the study who had baseline characteristics measured in each arm and overall.
Groups:
- Part 1A: FPA144 Dose Escalation Solid Tumors 1 mg/kg: 3 + 3 dose escalation cohort with 1.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1A: FPA144 Dose Escalation Solid Tumors 3 mg/kg: 3 + 3 dose escalation cohort with 3.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles..
- Part 1A: FPA144 Dose Escalation Solid Tumors 6 mg/kg: 3 + 3 dose escalation cohort with 6.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg: 3 + 3 dose escalation cohort with 10 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg: 3 + 3 dose escalation cohort with 15 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1B: FPA144 Dose Escalation Gastric 6 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 10 mg/kg IV every 2 weeks in 28 day cycles.
- Part 1B: FPA144 Dose Escalation Gastric 10 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 15 mg/kg IV every 2 weeks in 28 day cycles.
- Total: Total of all reporting groups
Arm/Group | Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 1 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 6 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 3 mg/kg | Part 1B: FPA144 Dose Escalation Gastric 6 mg/kg | Part 1B: FPA144 Dose Escalation Gastric 10 mg/kg | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 1 | 1 | 6 | 52 | 79
Age, Customized [Median (Full Range); unit: years] | 74 [39 to 76] | 64.5 [37 to 68] | 63 [52 to 75] | 62 [47 to 77] | 64 [61 to 80] | 59 [32 to 86] | 54 [54 to 54] | 39 [39 to 39] | 52 [40 to 65] | 57 [25 to 78] | 59 [25 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 | 2 | 2 | 1 | 0 | 3 | 21 | 33
  Male | 2 | 2 | 3 | 2 | 1 | 1 | 0 | 1 | 3 | 31 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 39 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 4 | 3 | 3 | 3 | 3 | 0 | 0 | 1 | 11 | 31
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 33 | 40
  United States | 3 | 4 | 3 | 3 | 3 | 3 | 0 | 0 | 1 | 14 | 34
  Taiwan | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Protocol Specified Dose-limiting Toxicities (Part 1 Only).
Description: Number of participants with grade 3 and grade 4 adverse events (AE) and clinical laboratory abnormalities defined as dose limiting toxicities (DLTs)
Time Frame: 4 weeks on average
Population: All patients who received FPA144
Measure: Count of Participants; unit: Participants
Groups:
- Part 1B: FPA144 Dose Escalation Gastric Cancer 3mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 3.0 mg/kg IV every 2 weeks in 28 day cycles.
- Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 6.0 mg/kg IV every 2 weeks in 28 day cycles.
- Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 10 mg/kg IV every 2 weeks in 28 day cycles.
Arm/Group | Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 1 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 6 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 3mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 1 | 1 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With AEs and Clinical Laboratory Abnormalities (Parts 1B and 2 Only)
Description: Number of Participants with AEs and clinical laboratory abnormalities (Parts 1B and 2 only)
Time Frame: 16 weeks on average
Population: All patients who received FPA144
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B: FPA144 Dose Escalation Gastric Cancer 3mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors
Number analyzed (Participants) | 1 | 1 | 6 | 52
Participants | 1 | 1 | 6 | 48

3. Secondary Outcome: Pharmacokinetic (PK) Profile of FPA144: Maximum Serum Concentration
Description: Sampling following the first dose in Part 1, pre and post-dose at selected cycles, and at the end of treatment for both Part 1 and Part 2.
  • Summary of area under serum concentration-time curve, maximum serum concentration,
Time Frame: 16 weeks on average
Population: All patients in the PK Full Analysis Population who have sufficient PK samples for the calculation of at least one PK parameter on at least one Study Day. Dose normalized PK parameters were reported so that patients at 0.3 mg/kg were excluded from mean value for part 1a because it is in the non-linear dose range.
Measure: Mean (Standard Deviation); unit: ug/ml
Groups:
- Phase 1a Dose Escalation 0.3 mg/kg: 3 + 3 dose escalation cohort with 0.3 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Phase 1a Dose Escalation 1 mg/kg: 3 + 3 dose escalation cohort with 1.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Phase 1a Dose Escalation 3 mg/kg: 3 + 3 dose escalation cohort with 3.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Phase 1a Dose Escalation 6 mg/kg: 3 + 3 dose escalation cohort with 6.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Phase 1a Dose Escalation 10 mg/kg: 3 + 3 dose escalation cohort with 10 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Phase 1a Dose Escalation 15 mg/kg: 3 + 3 dose escalation cohort with 15 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Phase 1b Dose Escalation in Gastric Cancer 3 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 3.0 mg/kg IV every 2 weeks in 28 day cycles.
- Phase 1b Dose Escalation in Gastric Cancer 6 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 6.0 mg/kg IV every 2 weeks in 28 day cycles.
- Phase 1b Dose Escalation in Gastric Cancer 10 mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 10 mg/kg IV every 2 weeks in 28 day cycles.
Arm/Group | Phase 1a Dose Escalation 0.3 mg/kg | Phase 1a Dose Escalation 1 mg/kg | Phase 1a Dose Escalation 3 mg/kg | Phase 1a Dose Escalation 6 mg/kg | Phase 1a Dose Escalation 10 mg/kg | Phase 1a Dose Escalation 15 mg/kg | Phase 1b Dose Escalation in Gastric Cancer 3 mg/kg | Phase 1b Dose Escalation in Gastric Cancer 6 mg/kg | Phase 1b Dose Escalation in Gastric Cancer 10 mg/kg | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors
Number analyzed (Participants) | 0 | 4 | 3 | 3 | 3 | 3 | 1 | 1 | 5 | 49
ug/ml |  | 0.2483 (0.08763) | 0.3117 (0.06536) | 0.2873 (0.02793) | 0.4097 (0.03208) | 0.3847 (0.14931) | 0.4900 (0) | 0.232 (0) | 0.2990 (0.06690) | 0.3145 (0.06981)

4. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 16 weeks on average
Population: Patients with various levels of FGFR2b overexpression in tumor samples treated with bemarituzumab who had baseline and post baseline scans performed.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1A: FPA144 Dose Escalation Solid Tumors 1.0 mg/kg: 3 + 3 dose escalation cohort with 1.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1A: FPA144 Dose Escalation Solid Tumors 3.0 mg/kg: 3 + 3 dose escalation cohort with 3.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1A: FPA144 Dose Escalation Solid Tumors 6.0 mg/kg: 3 + 3 dose escalation cohort with 6.0 mg/kg FPA144 IV every 2 weeks in 28 day cycles.
- Part 1B: FPA144 Dose Escalation Gastric Cancer 6mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 6.0 mg/kg IV every 2 weeks in 28 day cycles.
- Part 1B: FPA144 Dose Escalation Gastric Cancer 10mg/kg: 3 + 3 dose escalation cohort with expansion enrolling patients with gastric cancer. Tumors tested retrospectively for FGFR2 gene-amplified or FGFR2b protein-overexpressed. Expansion patients enrolled at dose levels cleared in Part 1A. Patients administered FPA144 10 mg/kg IV every 2 weeks in 28 day cycles.
Arm/Group | Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 1.0 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 3.0 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 6.0 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 3mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 6mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 10mg/kg | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 3 | 3 | 1 | 1 | 6 | 49
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4

5. Secondary Outcome: Duration of Response Per RECIST 1.1 (Part 2 Only)
Description: Duration of complete or partial response with 95% confidence intervals in gastric cancer population.
Time Frame: 16 weeks on average
Population: Gastric cancer patients with various levels of FGFR2b overexpression treated with FPA144 who had an objective response.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Part 1/2: FPA144 Dose Expansion Gastric or Other Solid Tumors: Gastric and bladder cancer patients with tumors with FGFR2b overexpression administered FPA144 15mg/kg IV every 2 weeks in 28 day cycles. Dose established from prior dose escalation evaluation in parts 1A and 1B.
Arm/Group | Part 1/2: FPA144 Dose Expansion Gastric or Other Solid Tumors
Number analyzed (Participants) | 6
Weeks | 14.1 [9.1 to 19.1]

6. Secondary Outcome: Pharmacokinetic (PK) Profile of FPA144: Area Under Serum Concentration-time Curve
Description: as for outcome 3
Time Frame: 16 weeks on average
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ug*day/ml
Arm/Group | Phase 1a Dose Escalation 0.3 mg/kg | Phase 1a Dose Escalation 1 mg/kg | Phase 1a Dose Escalation 3 mg/kg | Phase 1a Dose Escalation 6 mg/kg | Phase 1a Dose Escalation 10 mg/kg | Phase 1a Dose Escalation 15 mg/kg | Phase 1b Dose Escalation in Gastric Cancer 3 mg/kg | Phase 1b Dose Escalation in Gastric Cancer 6 mg/kg | Phase 1b Dose Escalation in Gastric Cancer 10 mg/kg | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors
Number analyzed (Participants) | 0 | 4 | 3 | 3 | 3 | 3 | 1 | 1 | 3 | 49
ug*day/ml |  | 1.288 (0.5159) | 1.547 (0.2902) | 1.427 (0.2367) | 1.863 (0.4119) | 1.697 (0.1464) | 2.69 (0) | 1.59 (0) | 1.648 (0.4055) | 1.867 (0.4495)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Cycle 1 Day 1 through completion of End-of-Treatment visit or until 28 days after last dose of study drug was administered.
Groups:
- Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg: 3 + 3 dose escalation cohort with 15mg/kg FPA144 IV every 2 weeks in 28 day cycles.
Arm/Group | Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 1.0 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 3.0 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 6.0 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg | Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 3 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg | Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/3 | 0/3 | 0/3 | 0/3 | 0/1 | 0/1 | 0/6 | 5/52
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4 | 2/3 | 0/3 | 0/3 | 1/3 | 0/1 | 0/1 | 2/6 | 17/52
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 3/3 | 2/3 | 3/3 | 1/1 | 1/1 | 6/6 | 48/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 1.0 mg/kg (N=4) | Part 1A: FPA144 Dose Escalation Solid Tumors 3.0 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 6.0 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg (N=3) | Part 1B: FPA144 Dose Escalation Gastric Cancer 3 mg/kg (N=1) | Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg (N=1) | Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg (N=6) | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors (N=52)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain, Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limbal stem cell deficiency (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoas Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Azotemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corneal Dystrophy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Device Malfunction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: FPA144 Dose Escalation Solid Tumors 0.3 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 1.0 mg/kg (N=4) | Part 1A: FPA144 Dose Escalation Solid Tumors 3.0 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 6.0 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 10 mg/kg (N=3) | Part 1A: FPA144 Dose Escalation Solid Tumors 15 mg/kg (N=3) | Part 1B: FPA144 Dose Escalation Gastric Cancer 3 mg/kg (N=1) | Part 1B: FPA144 Dose Escalation Gastric Cancer 6 mg/kg (N=1) | Part 1B: FPA144 Dose Escalation Gastric Cancer 10 mg/kg (N=6) | Part 2: FPA144 Dose Expansion Gastric or Other Solid Tumors (N=52)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 14
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eustachian Tube Obstruction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Eye (Eye disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 7
Eye Disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation Increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Limbal Stem Cell Deficiency (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metamorphosia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal Distention (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 8
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 14
Oesophageal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 7
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Early Satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 12
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 7
Anorectal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 4
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Weight Decreased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 16
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous System Disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystitis Non-infective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Operation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 14

LIMITATIONS AND CAVEATS:
Inclusion of patients with refractory gastric cancer with short duration of drug exposure may have limited our ability to accurately evaluate the incidence of off-target effects adverse events in the study population, in particular corneal toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT02318329/Prot_SAP_000.pdf